CLINICAL TRIAL: NCT00163319
Title: Comparison of Inhaled Ciclesonide (640 mcg/Day) and Fluticasone Propionate (1000 mcg/Day) in Patients With Moderate and Severe Persistent Asthma
Brief Title: Efficacy of Ciclesonide and Fluticasone Propionate in Adult Patients With Moderate and Severe Persistent Asthma (18 to 75 y) (BY9010/IT-101)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/IT-101
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Fluticasone propionate
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of the study is to compare the safety and efficacy of ciclesonide versus fluticasone propionate on the lung function, symptoms, use of rescue medication, and occurrence of side effects (such as candidiasis, hoarseness) in adults with persistent asthma. Ciclesonide will be inhaled twice daily at one dose level; fluticasone propionate will be inhaled twice daily at one dose level. The study duration consists of a baseline period (2 weeks) and a treatment period (24 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* History of bronchial asthma for at least 6 months
* Pre-treatment with CFC-beclomethasone dipropionate (CFC-BDP) ≥ 1000 mcg/day or equivalent and a long-acting beta agonist (LABA) either in free or fixed combination
* FEV1 ≥ 80% of predicted

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids or contraindications for the use of LABAs
* COPD
* Smoking with ≥10 pack-years
* Pregnancy
* Intention to become pregnant during the course of the study
* Breast feeding
* Lack of safe contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-11; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
number of patients with candidiasis of the oropharynx or hoarseness.

SECONDARY OUTCOMES:
inhaled Corticosteroids Questionnaire (ICQ)
proportion of cases of candidiasis of the oropharynx or
hoarseness at each visit Secondary variables
FEV1, FVC, PEF from spirometry
morning and evening PEF from diaries
diurnal PEF fluctuation
onset of treatment effect
percent days on which patient perceived asthma control
percent of nocturnal awakening-free days
percent of rescue medication free days
percent symptom free days
asthma symptom score
use of rescue medication
time to first asthma exacerbation
number of patients with an asthma exacerbation
AQLQ
number of patients with candidiasis of the oropharynx or hoarseness by severity
physical examination, ECG
vital sings
adverse events
standard laboratory work-up
morning serum cortisol
skin bruising.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (79):
- Belgium (8):
  - Altana Pharma/Nycomed, Brussels
  - Altana Pharma/Nycomed, Halen
  - Altana Pharma/Nycomed, Jette
  - Altana Pharma/Nycomed, Maison-Saint-Gérard
  - Altana Pharma/Nycomed, Namur
  - Altana Pharma/Nycomed, Ostend
  - Altana Pharma/Nycomed, Turnhout
  - Altana Pharma/Nycomed, Veurne
- France (15):
  - Altana Pharma/Nycomed, Aix-en-Provence
  - Altana Pharma/Nycomed, Béziers
  - Altana Pharma/Nycomed, Chauny
  - Altana Pharma/Nycomed, Grasse
  - Altana Pharma/Nycomed, La Rochelle
  - Altana Pharma/Nycomed, Marseille
  - Altana Pharma/Nycomed, Martigues
  - Altana Pharma/Nycomed, Metz
  - Altana Pharma/Nycomed, Montfermeil
  - Altana Pharma/Nycomed, Montpellier
  - Altana Pharma/Nycomed, Nice
  - Altana Pharma/Nycomed, Nîmes
  - Altana Pharma/Nycomed, Paris
  - Altana Pharma/Nycomed, Perpignan
  - Altana Pharma/Nycomed, Vieux-Condé
- Italy (13):
  - Altana Pharma/Nycomed, Ancona
  - Altana Pharma/Nycomed, Brescia
  - Altana Pharma/Nycomed, Chieti
  - Altana Pharma/Nycomed, Florence
  - Altana Pharma/Nycomed, Livorno
  - Altana Pharma/Nycomed, Milan
  - Altana Pharma/Nycomed, Milazzo (ME)
  - Altana Pharma/Nycomed, Napoli
  - Altana Pharma/Nycomed, Pavia
  - Altana Pharma/Nycomed, Pirri-Cagliari
  - Altana Pharma/Nycomed, Pordenone
  - Altana Pharma/Nycomed, Roma
  - Altana Pharma/Nycomed, Verona
- Netherlands (8):
  - Altana Pharma/Nycomed, Almere Stad
  - Altana Pharma/Nycomed, Haarlem
  - Altana Pharma/Nycomed, Harderwijk
  - Altana Pharma/Nycomed, Heerlen
  - Altana Pharma/Nycomed, Helmond
  - Altana Pharma/Nycomed, Schiedam
  - Altana Pharma/Nycomed, Utrecht
  - Altana Pharma/Nycomed, Veldhoven
- Spain (9):
  - Altana Pharma/Nycomed, Almería
  - Altana Pharma/Nycomed, Barcelona
  - Altana Pharma/Nycomed, Córdoba
  - Altana Pharma/Nycomed, Elche
  - Altana Pharma/Nycomed, Guadalajara
  - Altana Pharma/Nycomed, Madrid
  - Altana Pharma/Nycomed, Requena
  - Altana Pharma/Nycomed, San Sebastián
  - Altana Pharma/Nycomed, Valencia
- Switzerland (10):
  - Altana Pharma/Nycomed, Basel
  - Altana Pharma/Nycomed, Bellinzona
  - Altana Pharma/Nycomed, Bern
  - Altana Pharma/Nycomed, Bruderholz
  - Altana Pharma/Nycomed, La Chauxe-de-Fonds
  - Altana Pharma/Nycomed, Lugano
  - Altana Pharma/Nycomed, Münchenstein
  - Altana Pharma/Nycomed, Münsingen
  - Altana Pharma/Nycomed, Münsterlingen
  - Altana Pharma/Nycomed, Zurich
- United Kingdom (16):
  - Altana Pharma/Nycomed, Belfast
  - Altana Pharma/Nycomed, Belfast, Irland
  - Altana Pharma/Nycomed, Bradford on Avon, Wiltshire
  - Altana Pharma/Nycomed, Chesterfield Derbyshire
  - Altana Pharma/Nycomed, Chippenham, Wiltshire
  - Altana Pharma/Nycomed, Co. Antrim
  - Altana Pharma/Nycomed, Downpatrick, Northern Ireland
  - Altana Pharma/Nycomed, Dronfield
  - Altana Pharma/Nycomed, Glengormley
  - Altana Pharma/Nycomed, Glengormley Newtownabbey
  - Altana Pharma/Nycomed, Hastings
  - Altana Pharma/Nycomed, Maidenhead, Berks
  - Altana Pharma/Nycomed, Nottingham
  - Altana Pharma/Nycomed, Solihull
  - Altana Pharma/Nycomed, Warminster Wiltshire
  - Altana Pharma/Nycomed, Watford

REFERENCES:
- See also: BY9010-IT-101-RDS-2006-09-21.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4510&filename=BY9010-IT-101-RDS-2006-09-21.pdf